CLINICAL TRIAL: NCT01605097
Title: High Dose Rate Prostate (HDR) Brachytherapy Dose Escalation to Dominant Intra-prostatic Nodule for Patients With Intermediate and High Risk Prostate Cancer
Brief Title: High Dose Rate Prostate Brachytherapy: Dose Escalation to Dominant Intra-prostatic Nodule
Acronym: Dosepainting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H12-00557
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: prostate neoplasms; interstitial radiation; High dose rate prostate brachytherapy; dose escalation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HDR interstitial brachytherapy (Experimental): HDR prostate brachytherapy with dose escalation to 1250 cGy to the MRI-defined dominant intraprostatic lesion
  Interventions: Radiation: HDR interstitial brachytherapy

INTERVENTIONS:
Radiation: HDR interstitial brachytherapy — 2 treatments of 1000 cGy will be delivered to the entire prostate volume while escalating the dose to the visible disease to 1250 cGy
  Other Names: Planning soft ware Varian Medical Systems Vitesse III

SUMMARY:
This study will investigate the feasibility of using technology of ultrasound guided HDR brachytherapy to focally increase dose to regions within the prostate that are heavily infiltrated with cancer. Such regions, referred to as dominant intraprostatic lesions (DIL) can be visualized using diffusion contrast enhanced MRI employing an endo-rectal coil. The magnetic resonance (MR) images can be fused with the planning transrectal ultrasound (TRUS) prior to the brachytherapy procedure to design a dose distribution that will encompass the malignant volume with higher than the prescription dose. By its nature, brachytherapy has subvolumes that receive (for example)125% of the prescription dose or 150% of the prescription dose. With TRUS-guided and TRUS-planned HDR these areas can be manipulated to coincide with the DIL. The limit of dose escalation has been reached at whole prostate external beam doses of 81-86 Gy and still failure rates for intermediate and high risk disease are unacceptable. There is much interest in focal dose escalation and TRUS-guided HDR brachytherapy is perfectly suited to achieving this.

DETAILED DESCRIPTION:
Methods: If a dominant nodule is visualized on dynamic contrast enhanced (DCE) MRI, it will be contoured in 3D and the images fused to the planning TRUS study that is done in preparation for brachytherapy (of any type: seeds or HDR). The patient's treatment will consist of the standard combined external beam (4600 centiGray (cGy) in 23 fractions) and HDR brachytherapy boost (2 fractions of 1000 cGy given on days 5 and 15 of the external beam course). During each HDR treatment the plan will be manipulated such that the normally occurring high dose regions (125%, 150%) are positioned at the site of the identified disease. Normally approximately 60% of the prostate volume receives 125% of the dose and 30% receives 150%. By ensuring that the inherent dosimetry favors treatment of the known cancer, no region of the prostate would be "underdosed". HDR treatments are performed under general anesthesia as an out patient procedure.

Statistical Analysis: This is a feasibility study and the data reported will be descriptive including the frequency with which the DIL can be visualized in this population, the DIL volume compared to total prostate volume, and the isodose that can encompass the DIL without violating dose constraints to adjacent organs (urethra and bladder). Toxicity will be monitored and efficacy will be assessed by repeat DCE MRI at 12 months and biopsy at 30 months.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven adenocarcinoma of the prostate
* intermediate or high risk prostate cancer

  * Intermediate risk prostate cancer patients must have:

    * Clinical stage ≤ T2c,
    * Gleason score = 7 and initial prostate specific antigen (iPSA) ≤ 20, or
    * Gleason score ≤ 6 and iPSA > 10 and ≤ 20.
  * High risk patients may have

    * Clinical stage T3
    * Gleason score 8-10
    * PSA > 20 ng/ml
* fit for general anesthetic.
* unilateral disease with either a palpable nodule or a cluster of positive biopsies from a single region suggesting the presence of dominant nodule.
* estimated life expectancy of at least 10 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
* no contraindications to interstitial prostate brachytherapy.
* if on coumadin therapy must be able to stop safely for 7 days.
* must not have any contraindications to MRI

Exclusion Criteria:

* Does not meet staging criteria for intermediate or high risk prostate cancer
* Does not have a localized high volume of intraprostatic disease
* unfit for general anesthetic
* MRI contraindicated
* unable to stop blood thinners
* Life expectancy < 10 years

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Schmid, MSc, Principal Investigator — Medical Physicst
Locations (1):
- Cancer Center for the Southern Interior, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Groenendaal G, van den Berg CA, Korporaal JG, Philippens ME, Luijten PR, van Vulpen M, van der Heide UA. Simultaneous MRI diffusion and perfusion imaging for tumor delineation in prostate cancer patients. Radiother Oncol. 2010 May;95(2):185-90. doi: 10.1016/j.radonc.2010.02.014. Epub 2010 Mar 16. PMID 20231041
- [Background] Kim Y, Hsu IC, Lessard E, Kurhanewicz J, Noworolski SM, Pouliot J. Class solution in inverse planned HDR prostate brachytherapy for dose escalation of DIL defined by combined MRI/MRSI. Radiother Oncol. 2008 Jul;88(1):148-55. doi: 10.1016/j.radonc.2007.11.024. Epub 2008 Feb 20. PMID 18083260
- [Background] Pouliot J, Kim Y, Lessard E, Hsu IC, Vigneron DB, Kurhanewicz J. Inverse planning for HDR prostate brachytherapy used to boost dominant intraprostatic lesions defined by magnetic resonance spectroscopy imaging. Int J Radiat Oncol Biol Phys. 2004 Jul 15;59(4):1196-207. doi: 10.1016/j.ijrobp.2004.02.055. PMID 15234056
- [Derived] De Bari B, Daidone A, Alongi F. Is high dose rate brachytherapy reliable and effective treatment for prostate cancer patients? A review of the literature. Crit Rev Oncol Hematol. 2015 Jun;94(3):360-70. doi: 10.1016/j.critrevonc.2015.02.003. Epub 2015 Feb 17. PMID 25819287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Aim of protocol was to have 25 patients for whom dominant lesion identified on MRI and dose escalation feasible with HDR brachytherapy
Pre-assignment Details: One patient consented but ineligible because did not have a visible lesion on the MRI of his prostate.
Groups:
- High Dose Rate (HDR) Interstitial Brachytherapy: HDR prostate brachytherapy with dose escalation to 1250 cGy to the MRI-defined dominant intraprostatic lesion
  HDR interstitial brachytherapy: 2 treatments of 1000 cGy will be delivered to the entire prostate volume while escalating the dose to the visible disease to 1250 cGy
Period: Overall Study
Arm/Group | High Dose Rate (HDR) Interstitial Brachytherapy
Started | 26 (One patient consented but was ineligible due to lack of lesion visible on mpMRI)
Completed | 25
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | HDR Interstitial Brachytherapy
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 63 [51 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Baseline PSA ng/mL [Median (Full Range); unit: ng/mL] — Prostate-specific antigen, or PSA, is a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA test measures the level of PSA in a man's blood. For this test, a blood sample is sent to a laboratory for analysis.
  ng/mL | 10.4 [3.0 to 20.0]
Gleason score [Number; unit: participants] — Gleason score is assigned by pathologist on examination of prostate biopsy material and ranges from 2 to 10 with higher score representing more aggressive undifferentiated tumors
  participants
    Gleason 7 | 23
    Gleason 8 or 9 | 2
clinical stage [Number; unit: participants] — Clinical Tumor Stage is assigned from combination of digital rectal exam and imaging. T1 representants tumor that is neither palpable nor visible on imaging. cT2a and cT2b represent palpable/visible disease that is either less than half of one lobe (cT2a) or more than half of one lobe(cT2b).
  participants
    Stage T1c | 3
    Stage T2a | 7
    Stage T2b | 15

OUTCOME MEASURES:

1. Primary Outcome: Average Mean Dose to 90% of DIL Volume
Description: Feasibility of dose escalation to a minimum dose of 125% of prescription to 90% of the dominant intra-porstatic lesion (DIL) volume as defined on multiparametric endo-rectal magnetic resonance imaging (mpMRI) without exceeding critical organ dose constraints (Urethral volume receiving 115%= 0, Dose to 1cc of rectal wall < 7 Gy). 2 Fractions were performed and the mean dose to 90% of DIL volume was averaged.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Grays
Groups:
- High Dose Rate (HDR) Interstitial Brachytherapy: HDR prostate brachytherapy with dose escalation to 1250 centiGray (cGy) to the MRI-defined dominant intraprostatic lesion
  HDR interstitial brachytherapy: 2 treatments of 1000 cGy will be delivered to the entire prostate volume while escalating the dose to the visible disease to 1250 cGy
Arm/Group | High Dose Rate (HDR) Interstitial Brachytherapy
Number analyzed (Participants) | 25
Grays | 13.25 (1.1)

2. Secondary Outcome: Acute Toxicity
Description: Time to normalize International Prostate Symptom Score (months). Score range 0-35 with 35 being worst outcome. Normalization refers to a return to baseline urinary function prior to treatment.
Time Frame: 24 months
Population: Months to normalization of International Prostate Symptom Score following treatment.
Measure: Median (Full Range); unit: months
Arm/Group | HDR Interstitial Brachytherapy
Number analyzed (Participants) | 25
months | 1.5 [0.6 to 9.0]

3. Secondary Outcome: Prostate Specific Antigen(PSA) Response at 5-years
Description: Efficacy assessed by biochemical PSA response reported at median 5 year follow up.
Time Frame: 5 years
Population: All 25 underwent dose escalation to dominant lesion in prostate to median 132% of prescription dose
Measure: Median (Full Range); unit: ng/ml
Arm/Group | HDR Interstitial Brachytherapy
Number analyzed (Participants) | 25
ng/ml | 0.06 [0.02 to 0.18]

ADVERSE EVENTS:
Time Frame: Data collected for 60 months on all patients. Accrual was completed July 2013 and data collected to July 2018.
Description: CTCAE V 3.0
Arm/Group | HDR Interstitial Brachytherapy
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDR Interstitial Brachytherapy (N=25)
late hematuria grade 1 (Renal and urinary disorders) | 2 (2)
grade 1 proctitis (Gastrointestinal disorders) | 3 (3) — rectal discomfort, no intervention required

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No